CLINICAL TRIAL: NCT01399762
Title: International Multicenter Registry for Mechanical Recanalization Procedures in Acute Stroke (ENDOSTROKE)
Brief Title: International Multicenter Registry for Mechanical Recanalization Procedures in Acute Stroke
Acronym: ENDOSTROKE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Goethe University (Other)
Responsible Party: PD Dr. med. Oliver C. Singer, Hirngefaesszentrum der Goethe Universitaet
Other Study IDs: Endostroke_01
Record Dates: First submitted 2011-07-18; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Acute Stroke
Keywords: stroke, acute; mechanical recanalization; interventional neuroradiology; clinical registry
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- mechanical recanalization: Patients with acute stroke being treated with endovascular devices for mechanical recanalization (no restriction to specific endovascular devices)
  Interventions: Device: mechanical recanalization

INTERVENTIONS:
Device: mechanical recanalization — Endovascular thrombus extraction by mechanical recanalization devices

SUMMARY:
The purpose of the Endostroke Registry is to gather information on predictors of good or poor clinical outcome following mechanical recanalization therapies for acute ischemic stroke.

DETAILED DESCRIPTION:
Mechanical recanalization procedures are increasingly used in large vessel stroke, i.e. in proximal middle cerebral artery (MCA) or basilar artery (BA) occlusion. This trend is due to the limited efficacy of the only approved acute stroke treatment, systemic thrombolysis, in large vessel occlusion but also due to new technical innovations triggering the development of numerous devices for thrombus extraction. Within large single-arm trials, some of these devices demonstrated their potential with respect to acceptable complication- and substantial recanalization rates. Nevertheless, clinical outcome of these stroke patients is frequently poor despite an elaborate, aggressive, but also complex and costly treatment regimen. The factors determining good or poor clinical outcome in mechanical recanalization remain to be determined. The goal of the ENDOSTROKE-registry is the systemic evaluation of technical and clinical features that might be important for the further development and evaluation of endovascular treatment strategies for acute stroke. Special emphasis is laid on the assessment of clinical outcome (90 day MRS). Concerning technical and periprocedural aspects, a focus is put on time issues i.e. intra-hospital time delays, duration of angiographic procedures until vessel patency is achieved.It is planned to enroll approximately 500 patients in this registry. In first line, prospective patients will be included in the register (start date January 2011) but retrospective inclusion of patients being treated within the three years before the start of the register is allowed as long a consecutive patient registration is guaranteed (to exclude selection bias). Data analysis will include univariate and multivariate approaches with respect to clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated with mechanical recanalization devices due to an acute proximal arterial vessel occlusion of brain supplying arteries

Exclusion Criteria:

* Patients being treated with mechanical recanalization devices for venous vessel occlusion.
* Patients being treated with mechanical recanalization devices due to an acute vessel occlusion which occured as a complication of an angiographic procedure scheduled for other reasons (i.e. as a complication of a diagnostic angiography or coiling procedure for cerebral aneurysms)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke being treated with mechanical recanalization devices for proximal vessel occlusion of brain supplying arteries (i.e. MCA main stem occlusion, basilar artery occlusion, distal ICA occlusion)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-01

PRIMARY OUTCOMES:
Clinical outcome | approx. 90 days after stroke onset
  Proportion of patients with favourable clinical outcome defined as a Modified Rankin Score (MRS) of 0,1, or 2 three months after the intervention.

SECONDARY OUTCOMES:
Angiographic outcome | Day of intervention
  Proportion of patients with complete recanalization defined as Thrombolysis in Myocardial Infarction (TIMI) Grade 2 or 3.
Complication rate | within 36 h after endovascular procedure
  Periprocedural complication rate defined as a combination of symptomatic intracranial hemorrhage (ECASS classification PH I and PH II), subarachnoid hemorrhage and thrombembolic events.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver C. Singer, MD, Principal Investigator — Hirngefaesszentrum Goethe University Frankfurt Germany; Joachim Berkefeld, MD, Principal Investigator — Hirngefaesszentrum Goethe University Frankfurt Germany
Locations (13):
- Austria (2):
  - Departments of Neurology and Neuroradiology, University Hospital, Graz
  - Departments of Neurology and Neuroradiology, Landes-Nervenklinik Wagner-Jauregg, Linz
- Germany (11):
  - Departments of Neurology and Neuroradiology, University Hospital, Aachen
  - Departments of Neurology and Radiology, Klinikum Altenburger Land, Altenburg
  - Departments of Neurology and Neuroradiology, Charite University Hospital, Berlin
  - Departments of Neurology and Neuroradiology, University Hospital, Düsseldorf
  - Departments of Neurology and Neuroradiology, University Hospital, Essen
  - Hirngefaesszentrum Goethe University, Frankfurt
  - Departments of Neurology and Neuroradiology, Klinikum Fulda, Fulda
  - Departments of Neurology and Neuroradiology, University Hospital, Giessen
  - Departments of Neurology and Neuroradiology, University Hospital, Kiel
  - Departments of Neurology and Neuroradiology, University Hospital, Mainz
  - Departments of Neurology and Neuroradiology, Knappschaftskrankenhaus, Recklinghausen